CLINICAL TRIAL: NCT07146594
Title: Clinical Evaluation of a 14day Modified Bismuth Quadruple Therapy for the Eradication of H. Pylori in a High Clarithromycin and Metronidazole Resistance Area
Brief Title: Clinical Evaluation of a 14day Modified Bismuth Quadruple Therapy for the Eradication of Helicobacter Pylori in a High Clarithromycin and Metronidazole Resistance Area Regarding Patients With Peptic Ulcer and Non Ulcer Dyspepsia
Acronym: MBISQ4HP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Athens Medical Center (Other)
Responsible Party: Principal Investigator, ILIAS XIROUCHAKIS, Dr Ilias Xirouchakis MD, FEBGH, Athens Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105/2005
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Helicobacter Pylori Gastritis; Helicobacter Eradication
Keywords: Helicobacter pylori eradication

STUDY DESIGN:
Intervention Model Description: Eligible patients of the study group will receive treatment whether as first line if no treatment for helicobacter pylori has been given before or rescue therapy if any other than the study treatment protocol has been given and failed to eradicate helicobacter pylori
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Helicobacter pylori infected (Active Comparator): This arm will include patients who have to receive eradication therapy for the first time as first line or experienced patients who have to receive eradication as rescue therapy for third or further line, respectively.
  Interventions: Drug: Modified bismuth-containing eradication treatment

INTERVENTIONS:
Drug: Modified bismuth-containing eradication treatment — After the confirmation of Helicobacter pylori infection, eligible patients whether first line or rescue therapy will be assigned to receive:
  - A modified and optimized bismuth quadruple therapy that comprises: 40 mg of esomeprazole bid, amoxicillin 1g tds, metronidazole 500mg tds and bismuth subcitrate 240mg bid, all medications taken for 14 days.
  Esomeprazole will be given at least 30 minutes before meals every 12 hours. Antibiotics will be given after meals every 8 hours and bismuth subcitrate at least 2 hours far from meals every 12 hours.

SUMMARY:
The goal of this clinical trial is to learn if a modified bismuth-containing therapy for the treatment of helicobacter pylori infection works to treat chronic helicobacter pylori related gastritis in adults treated either for first time or after a previous failure of another helicbacter erdication therapy. It will also learn about the safety and compliance of the modified bismuth containing therapy for helicobacter pylori.

The main questions it aims to answer are:

Does the modified bismuth-containing therapy for helicobacter pylori maintains a high eradication profile? What medical problems do participants have when taking the bismuth containing therapy? Researchers will present the eradication percentage of the modified bismuth containing therapy for helicobacter pylori in a difficult to treat population with a high profile of resistance to antibiotics for the treatment of helicobacter pylori separately for first time treated patients or patients with previous failures of other therapies.

Participants will:

Take the modified bismuth containing therapy which consists of four different medications (esomeprazole, amoxicillin, metronidazole, bismuth subcitrate) taken for 14 days in selected timepoints.

Visit the clinic at the end of therapy for checkups and at 6 to 8 weeks after the end of therapy for final evaluation of completed eradication.

Keep a diary of their symptoms and the number of medications taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years or older with dyspepsia or iron deficiency anaemia, referring for upper GI endoscopy and found to be infected with Helicobacter pylori (positive rapid urease test or histology), naïve or experienced to H. pylori eradication treatment, will be invited to participate in the study.

Exclusion Criteria:

* Exclusion criteria are: age below 18 years, presence of severe co-morbidities (i.e. liver cirrhosis, renal failure, haematological, neurological, psychiatric, severe cardiovascular or pulmonary disease), previous gastric surgery, gastric malignancies, Zollinger-Elisson syndrome, known allergy or other contraindications to the study medications, previous H. pylori bismuth containing therapies, use of antibiotics , bismuth salts , NSAIDS or aspirin in the preceding month, use of PPI in the preceding two weeks and not willing to participate in the study. Pregnant or lactating women will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness to eradicate helicobacter pylori with modified bismuth-containing treatment | From enrollment to the end of treatment and assessment of eradication results at 8-10 weeks
  Participants achieved helicobacter pylori eradication if they perform negative at 13C-urea breath test (13C-UBT) 6-8 weeks after completion of modified bismuth-containing treatment

SECONDARY OUTCOMES:
Secondary outcomes are to assess patient's compliance and adverse events | From enrollment to the end of evaluation at 8 weeks
  Side effects of treatment will be assessed on a structured clinical interview with a specific questionnaire completed immediately after the end of eradication therapy and at the final re-evaluation at 8 weeks. During the interview, patients will be asked to grade the severity of each adverse event experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with common everyday activities), or "severe" (causing considerable interference with patients' daily activities). Incapacitating or life-threatening complications will be classified as serious and will be reported to regulatory agency (National Organization of Medicines). Adherence to treatment will be assessed by providing all patients with a pre-structured printed table with all dosages illustrated, asking to tick each time a pill was consumed and bring it back along with any tablet not consumed, for pill counting.

OTHER OUTCOMES:
Other outcome is to assess patient's compliance rescue therapies performance according to resistance profile. | From enrollment to evaluation at 8 weeks
  In patients that are eligible to receive a rescue therapy, H. pylori clinical strains will be isolated from gastric biopsies. Antibiotic susceptibility testing of Helicobacter pylori will be performed utilizing E-test strips (BioMerieux, Marcy l'Étoile, France), according to the manufacturer's instructions, on Mueller Hinton agar medium (Beckton Dickinson) supplemented with 10% horse blood. MIC clinical breakpoints used to define resistance according to EUCAST will be: clarithromycin (>0.5 mg/L), levofloxacin (>1 mg/L), tetracycline (>1 mg/L), metronidazole (>8 mg/L) and amoxicillin (>0.12 mg/L).

REFERENCES:
- [Background] Graham DY, Dore MP, Lu H. Understanding treatment guidelines with bismuth and non-bismuth quadruple Helicobacter pylori eradication therapies. Expert Rev Anti Infect Ther. 2018 Sep;16(9):679-687. doi: 10.1080/14787210.2018.1511427. Epub 2018 Aug 23. PMID 30102559
- [Background] Han Z, Li Y, Kong Q, Liu J, Wang J, Wan M, Lin M, Lin B, Zhang W, Ding Y, Wang S, Mu Y, Duan M, Zuo X, Li YQ. Efficacy of bismuth for antibiotic-resistant Helicobacter pylori strains eradication: A systematic review and meta-analysis. Helicobacter. 2022 Dec;27(6):e12930. doi: 10.1111/hel.12930. Epub 2022 Sep 25. PMID 36156332
- [Background] Megraud F. The challenge of Helicobacter pylori resistance to antibiotics: the comeback of bismuth-based quadruple therapy. Therap Adv Gastroenterol. 2012 Mar;5(2):103-9. doi: 10.1177/1756283X11432492. PMID 22423259
- [Background] Tsay FW, Wu DC, Yu HC, Kao SS, Lin KH, Cheng JS, Wang HM, Chen WC, Sun WC, Tsai KW, Hsu PI. A Randomized Controlled Trial Shows that both 14-Day Hybrid and Bismuth Quadruple Therapies Cure Most Patients with Helicobacter pylori Infection in Populations with Moderate Antibiotic Resistance. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e00140-17. doi: 10.1128/AAC.00140-17. Print 2017 Nov. PMID 28807915
- [Background] Georgopoulos SD, Xirouchakis E, Liatsos C, Apostolopoulos P, Kasapidis P, Martinez-Gonzalez B, Laoudi F, Stoupaki M, Axiaris G, Sgouras D, Mentis A, Michopoulos S. Equivalence Trial of the Non-Bismuth 10-Day Concomitant and 14-Day Hybrid Therapies for Helicobacter pylori Eradication in High Clarithromycin Resistance Areas. Antibiotics (Basel). 2024 Mar 20;13(3):280. doi: 10.3390/antibiotics13030280. PMID 38534715
- [Background] Georgopoulos SD, Xirouchakis E, Martinez-Gonzales B, Zampeli E, Grivas E, Spiliadi C, Sotiropoulou M, Petraki K, Zografos K, Laoudi F, Sgouras D, Mentis A, Kasapidis P, Michopoulos S. Randomized clinical trial comparing ten day concomitant and sequential therapies for Helicobacter pylori eradication in a high clarithromycin resistance area. Eur J Intern Med. 2016 Jul;32:84-90. doi: 10.1016/j.ejim.2016.04.011. Epub 2016 Apr 28. PMID 27134145
- [Background] Olmedo L, Calvet X, Gene E, Bordin DS, Voynovan I, Castro-Fernandez M, Pabon-Carrasco M, Keco-Huerga A, Perez-Aisa A, Lucendo AJ, Rodrigo L, Sarsenbaeva AS, Khlinov IB, Fadieienko G, Zaytsev O, Lanas A, Martinez-Dominguez SJ, Alfaro E, Jonaitis L, Nunez O, Pellicano R, Hernandez L, Gridnyev O, Kupcinskas J, Gasbarrini A, Boltin D, Niv Y, Babayeva G, Marcos-Pinto R, Tepes B, Venerito M, Papp V, Lerang F, Leja M, Phull PS, Marlicz W, Doulberis M, Smith SM, Milivojevic V, Kunovsky L, Mestrovic A, Matysiak-Budnik T, Simsek H, Cano-Catala A, Puig I, Moreira L, Parra P, Nyssen OP, Megraud F, O'Morain C, Gisbert JP; Hp-EuReg investigators*. Evolution of the use, effectiveness and safety of bismuth-containing quadruple therapy for Helicobacter pylori infection between 2013 and 2021: results from the European registry on H. pylori management (Hp-EuReg). Gut. 2024 Dec 10;74(1):15-25. doi: 10.1136/gutjnl-2024-332804. PMID 39461739
- [Background] Rokkas T, Gisbert JP, Malfertheiner P, Niv Y, Gasbarrini A, Leja M, Megraud F, O'Morain C, Graham DY. Comparative Effectiveness of Multiple Different First-Line Treatment Regimens for Helicobacter pylori Infection: A Network Meta-analysis. Gastroenterology. 2021 Aug;161(2):495-507.e4. doi: 10.1053/j.gastro.2021.04.012. Epub 2021 Apr 8. PMID 33839101
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Chen Q, Long X, Ji Y, Liang X, Li D, Gao H, Xu B, Liu M, Chen Y, Sun Y, Zhao Y, Xu G, Song Y, Yu L, Zhang W, Liu W, Graham DY, Lu H. Randomised controlled trial: susceptibility-guided therapy versus empiric bismuth quadruple therapy for first-line Helicobacter pylori treatment. Aliment Pharmacol Ther. 2019 Jun;49(11):1385-1394. doi: 10.1111/apt.15273. Epub 2019 Apr 24. PMID 31020673